CLINICAL TRIAL: NCT05110625
Title: Development and Evaluation of a Low Intensity, Multifaceted, Digital Health Intervention to Prevent Type 2 Diabetes Mellitus in the Primary Care Setting: the PREDIABETEXT Study
Brief Title: mHealth Intervention to Prevent Type 2 Diabetes Mellitus (Phase II Study)
Acronym: preDIABETEXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació d'investigació Sanitària de les Illes Balears (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SYN20/04
Record Dates: First submitted 2021-10-05; First posted 2021-11-08 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2022-08

CONDITIONS: Prediabetic State
Keywords: Prediabetic State; Glycemic Control; Telemedicine
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention A (Experimental): Participants will receive Messaging Intervention
  Interventions: Behavioral: preDIABE-TEXT
- Intervention B (Experimental): Participants will receive messaging intervention plus online education to their primary healthcare workers
  Interventions: Behavioral: preDIABE-TEXT; Other: Online Education
- Control (No Intervention): Participants will receive usual care only, and their healthcare workers will not receive online education

INTERVENTIONS:
Behavioral: preDIABE-TEXT — Participants will receive text messages (three per week) in their mobile phones during six months.
  Arms: Intervention A; Intervention B
Other: Online Education — Primary healthcare workers will receive an online educacion about prediabetes. This intervention will aim at: 1) raising awareness about the importance of T2DM prevention; 2) increasing knowledge about effective strategies for diabetes prevention; 3) improving knowledge about brief counselling techniques; and, 4) enhancing communication skills.
  Arms: Intervention B

SUMMARY:
The aim of this study is to develop and evaluate a low intensity, multifaceted, digital health intervention to prevent T2DM based on: i) the use of a system comprising mobile health (mHealth) technology integrated with electronic health records to send tailored text messages (SMSs) promoting lifestyle changes in people at risk of T2DM, and, ii) the provision of online education to primary healthcare workers about prediabetes management.

DETAILED DESCRIPTION:
The PREDIABETEXT project will involve five WorkPackages (WP). In WP1-4 we will develop and pilot-test the different components of the intervention (WP1 will develop the brief text messages targeted to patients; WP2 will adapt our existing technology system to deliver the messages; WP3 will develop an educational intervention targeted to Primary Healthcare workers, and; WP4 will pilot-test and optimise both interventions). In WP5 we will conduct a phase II, six-month, three-arm, cluster randomised, clinical trial with 42 primary care workers and 420 patients at risk of T2DM (HbA1c from 6% to 6.4% or fasting plasma glucose 110-125mg/dl, or both) registered in Primary Care centres from Mallorca. Patients will be allocated to a control (usual care) group, intervention A (patient messaging intervention), or intervention B (patient messaging intervention plus online education to their primary healthcare workers). The primary outcome will be HbA1c. Secondary outcomes will include additional clinical outcomes, and physiological, behavioural and psychological outcomes.

ELIGIBILITY:
ELIGIBILITY CRITERIA FOR PRIMARY HEALTHCARE WORKERS:

We will include physicians and nurses from primary care centres in Mallorca. We will exclude those anticipating moving to a different centre during the study period.

ELIGIBILITY CRITERIA FOR PATIENTS:

Inclusion Criteria:

* Registered in the Public Health Service of the Balearic Islands
* At risk of T2DM (HbA1c from 6% to 6.4% within the last 3 months or two consecutive values of fasting plasma glucose 110-125mg/dl within the last 12 months, or both)
* With access to a mobile device able to receive text messages.

Exclusion Criteria:

* People not able to read messages in Spanish
* Patients with severe mental conditions.
* Patients on an antidiabetic medication regime
* Pregnancy: currently or during the previous 12 months
* People planning to change healthcare centre during the intervention period

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Glycated Hemoglobin (HbA1C) at 6 months | Baseline and Postintervention (6 months)

SECONDARY OUTCOMES:
Change from Baseline Fasting blood glucose at 6 months | Baseline and Postintervention (6 months)
Change from Baseline Triglycerides at 6 months | Baseline and Postintervention (6 months)
Change from Baseline Total Cholesterol at 6 months | Baseline and Postintervention (6 months)
Change from Baseline low density cholesterol (LDL) at 6 months | Baseline and Postintervention (6 months)
Change from Baseline high density cholesterol (HDL) at 6 months | Baseline and Postintervention (6 months)
Change from Baseline lipoprotein A at 6 months | Baseline and Postintervention (6 months)
Change from Baseline aspartate aminotransferase enzyme (AST) at 6 months | Baseline and Postintervention (6 months)
Change from Baseline alanine aminotransferase (ALT) at 6 months | Baseline and Postintervention (6 months)
Change from Baseline gamma glutamil transpeptidase (GGT) at 6 months | Baseline and Postintervention (6 months)
Change from Baseline complete hemogram at 6 months | Baseline and Postintervention (6 months)
Change from Baseline creatinine at 6 months | Baseline and Postintervention (6 months)
Change from Baseline serum albumin at 6 months | Baseline and Postintervention (6 months)
Change from Baseline insuline at 6 months | Baseline and Postintervention (6 months)
Change from Baseline urinary sediment at 6 months | Baseline and Postintervention (6 months)
Change from Baseline albumin-craetinine ratio at 6 months | Baseline and Postintervention (6 months)
Change from Baseline Body Weight at 6 months | Baseline and Postintervention (6 months)
Change from Baseline Waist Circumference at 6 months | Baseline and Postintervention (6 months)
Change from Baseline Blood Pressure at 6 months | Baseline and Postintervention (6 months)
Change from Baseline of Cardiovascular disease risk at 6 months | Baseline and Postintervention (6 months)
  Cardiovascular disease risk determined using the REGICOR calculator (www.imim.cat; Ramos et al., 2003)
Diagnosis of T2DM | Postintervention (6 months)
Brief motivation questionnaire (ad hoc) | Baseline and Postintervention (6 months)
  On a scale from 0 to 7, this questionnaire meassures the level of motivation that participants present for following a healthy diet and a physical activity plan.
14-point Mediterranean diet adherence screener (MEDAS-14) | Baseline and Postintervention (6 months)
  Adherence to healthy diet. The score ranges from 0 to 14. A higher score corresponds to a higher adherence to Mediterranean diet. We will classify participants as low adherents (≤5), moderate adherents (6-9) or high adherents (≥10).
REGICOR Short form Physical Activity Questionnaire | Baseline and Postintervention (6 months)
  The questionnaire is a reliable and valid method to estimate moderate and vigorous intensity leisure time physical activity and sensitive to detect changes in moderate and vigorous intensity leisure time physical activity https://regicor.cat/aplicacions/activitat-fisica/
Spanish version of the physical activity questionnaire used in the Physical activity questionnaire from the Nurses' Health Study | Baseline and Postintervention (6 months)
  We will use the second part of the questionnaire, which studies sedentary behaviour. It includes questions about the number of hours spent in sedentary activities.
  Public Health Nutrition: 8(7), 920-927 https://nurseshealthstudy.org/
Global Adult Tobbacco Survey: GATS questionnaire. | Baseline and Postintervention (6 months)
  Tobbacco consumption. 3-items adapted from the GATS questionnaire (WHO).
Quantification of alcohol consumption - FISTERRA | Baseline and Postintervention (6 months)
  Calcultaion of alcohol consumption in Spanish Standard Drink units (10g per unit) per week.
  https://www.fisterra.com/herramientas/calcumed/

OTHER OUTCOMES:
Number of eligible patients | Baseline
Recruitment rate | Baseline
  follow-up rate
Follow-up rate | Postintervention (6 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Ignacio Ricci-Cabello, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Yes
We will share all collected IPD after anonymization
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available from January 2023 onwards
Access Criteria: Upon a reasonable request, we will grant access to public organizations. The PI of the project will review the requests.

REFERENCES:
- [Background] Soriguer F, Goday A, Bosch-Comas A, Bordiu E, Calle-Pascual A, Carmena R, Casamitjana R, Castano L, Castell C, Catala M, Delgado E, Franch J, Gaztambide S, Girbes J, Gomis R, Gutierrez G, Lopez-Alba A, Martinez-Larrad MT, Menendez E, Mora-Peces I, Ortega E, Pascual-Manich G, Rojo-Martinez G, Serrano-Rios M, Valdes S, Vazquez JA, Vendrell J. Prevalence of diabetes mellitus and impaired glucose regulation in Spain: the Di@bet.es Study. Diabetologia. 2012 Jan;55(1):88-93. doi: 10.1007/s00125-011-2336-9. Epub 2011 Oct 11. PMID 21987347
- [Background] Chow CK, Redfern J, Hillis GS, Thakkar J, Santo K, Hackett ML, Jan S, Graves N, de Keizer L, Barry T, Bompoint S, Stepien S, Whittaker R, Rodgers A, Thiagalingam A. Effect of Lifestyle-Focused Text Messaging on Risk Factor Modification in Patients With Coronary Heart Disease: A Randomized Clinical Trial. JAMA. 2015 Sep 22-29;314(12):1255-63. doi: 10.1001/jama.2015.10945. PMID 26393848
- [Derived] Mira-Martinez S, Malih N, Angullo-Martinez E, Zamanillo-Campos R, Yanez AM, Bennasar-Veny M, Gomez-Juanes R, Konieczna J, Jimenez R, Serrano-Ripoll MJ, Fiol-deRoque MA, Leiva A, Galmes-Panades AM, Miralles-Xamena J, Vidal-Thomas MC, Gomez-Cobo C, Gervilla E, Ona-Gil JI, Ricci-Cabello I. A Multifaceted Digital Intervention for the Prevention of Type 2 Diabetes Mellitus in Primary Care (PREDIABETEXT): Cluster Randomized Trial. J Med Internet Res. 2025 Oct 9;27:e70981. doi: 10.2196/70981. PMID 41067715